CLINICAL TRIAL: NCT03812198
Title: A Phase 1, 3-part, Single (Open-label) and Multiple (Double-blind, Placebo-controlled) Oral Dose Trial to Evaluate the Safety, Tolerability, and Pharmacokinetics of LEO 32731 Formulations in Healthy Subjects
Brief Title: A Trial to Investigate the Safety, Tolerability, and Drug Levels in Blood After Single and Multiple Doses of LEO 32731 in Healthy People
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: LP0058-1442; 2018-003282-34 (EudraCT Number)
Record Dates: First submitted 2019-01-18; First posted 2019-01-23 (Actual); Last update posted 2019-07-01 (Actual); Status verified 2019-06

CONDITIONS: Healthy
Keywords: healthy
MeSH Terms: interventions — Hardness

STUDY DESIGN:
Intervention Model Description: Part 1 (single dose, cross-over) Part 2 (single dose, cross-over with food effect evaluation) Part 3 (multiple dose, parallel)
Who Masked: Participant, Care Provider, Investigator
Masking Description: 3-part, single (open-label) and multiple (double-blind, placebo-controlled)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Group 1-1 (Active Comparator): Part 1: Subjects will receive 3 doses of LEO 32731 in different formulations, as follows (1 dose per formulation/treatment period): LEO 32731 modified release tablet; LEO 32731 blend, hard capsule; LEO 32731 API hard capsule (reference formulation).
  Interventions: Drug: LEO 32731 modified release tablet; Drug: LEO 32731 blend, hard capsule; Drug: LEO 32731 API, hard capsule
- Group 1-2 (Active Comparator): Part 1: Subjects will receive 3 doses of LEO 32731 in different formulations, as follows (1 dose per formulation/treatment period): LEO 32731 soft capsule; LEO 32731 gastro-resistant capsule; LEO 32731 API hard capsule (reference formulation).
  Interventions: Drug: LEO 32731 API, hard capsule; Drug: LEO 32731 soft capsule; Drug: LEO 32731 gastro-resistant capsule
- Group 2-1 (Experimental): Part 2: Subjects will receive 3 doses of the same LEO 32731 formulation under different conditions, as follow (1 dose per condition/treatment period): fasted, after low-fat breakfast, after high-fat breakfast.
  The formulation depends on the outcome of Part 1.
  Interventions: Drug: LEO 32731
- Group 2-2 (Experimental): Part 2: Subjects will receive 3 doses of the same LEO 32731 formulation under different conditions, as follow (1 dose per condition/treatment period): fasted, after low-fat breakfast, after high-fat breakfast.
  The formulation depends on the outcome of Part 1.
  Interventions: Drug: LEO 32731
- Group 2-3 (Experimental): Part 2: Subjects will receive 3 doses of the same LEO 32731 formulation under different conditions, as follow (1 dose per condition/treatment period): fasted, after low-fat breakfast, after high-fat breakfast.
  The formulation depends on the outcome of Part 1.
  Interventions: Drug: LEO 32731
- Group 3-1 (Placebo Comparator): Subjects will be dosed twice daily from Days 1-17 (morning dose only on Day 17) with LEO 32731 or placebo. The formulation depends on the outcome of Part 2.
  Interventions: Drug: LEO 32731; Other: Placebo
- Group 3-2 (Placebo Comparator): Subjects will be dosed twice daily from Days 1-17 (morning dose only on Day 17) with LEO 32731 or placebo. The formulation depends on the outcome of Part 2.
  Interventions: Drug: LEO 32731; Other: Placebo

INTERVENTIONS:
Drug: LEO 32731 modified release tablet — At each dosing, subjects will swallow the appropriate number of tablets with approximately 240 mL of water at room temperature.
  Arms: Group 1-1
Drug: LEO 32731 blend, hard capsule — At each dosing, subjects will swallow the appropriate number of capsules with approximately 240 mL of water at room temperature.
  Arms: Group 1-1
Drug: LEO 32731 API, hard capsule — At each dosing, subjects will swallow the appropriate number of capsules with approximately 240 mL of water at room temperature.
  Arms: Group 1-1; Group 1-2
Drug: LEO 32731 soft capsule — At each dosing, subjects will swallow the appropriate number of capsules with approximately 240 mL of water at room temperature.
  Arms: Group 1-2
Drug: LEO 32731 gastro-resistant capsule — At each dosing, subjects will swallow the appropriate number of capsules with approximately 240 mL of water at room temperature.
  Arms: Group 1-2
Drug: LEO 32731 — At each dosing, subjects will swallow the appropriate number of tablets or capsules with approximately 240 mL of water at room temperature.
  Arms: Group 2-1; Group 2-2; Group 2-3; Group 3-1; Group 3-2
Other: Placebo — At each dosing, subjects will swallow the appropriate number of tablets or capsules with approximately 240 mL of water at room temperature.
  Arms: Group 3-1; Group 3-2

SUMMARY:
This is a phase 1 trial to evaluate the safety, tolerability, and pharmacokinetics of 4 different oral formulations of LEO 32731 in healthy subjects. The trial will be conducted in 3 parts at a single site. Each eligible subject will be enrolled into 1 group only and will participate in 3 treatment periods.

DETAILED DESCRIPTION:
Part 1 will evaluate the pharmacokinetics of single doses of 4 test formulations of LEO 32731 compared with a reference formulation. Part 2 will evaluate the effect of food on the pharmacokinetics of selected test formulations of LEO 32731. Part 3 will evaluate the tolerability and safety of selected test formulations of LEO 32731 after multiple dosing.

Based on data from Part 1, up to 3 formulations will be taken forward to Part 2. If none of the formulations are considered appropriate to take forward to Part 2, the trial will stop after Part 1. Similarly, based on data from Part 2, up to 2 formulations will be taken forward to Part 3. If none of the formulations are considered appropriate to take forward to Part 3, the trial will stop after Part 2.

ELIGIBILITY:
Key inclusion criteria:

* Age 18 to 65 years, inclusive.
* Body mass index of 18.5 to 29.9 kg/m2, inclusive.
* In good health, at the discretion of the investigator, as determined by: medical history, physical examination, vital sign assessment (specifically, blood pressure must be within normal reference range), 12-lead ECG, clinical laboratory evaluations, aspartate aminotransferase and alanine aminotransferase not above the upper limit of normal (Gilbert's syndrome is not acceptable).
* Female subjects of childbearing potential must be willing to use a highly effective form of birth control in conjunction with a barrier method of contraception throughout the trial and for at least 90 days after final follow-up.
* Male subjects with a female partner of childbearing potential must be willing to use a highly effective form of birth control in conjunction with male barrier method of contraception (i.e. male condom with spermicide) throughout the trial and for at least 90 days after final follow-up.

Key exclusion criteria:

* Systemic or topical treatment within 14 days prior to first dose administration unless in the opinion of the investigator the medication will not interfere with the trial procedures or compromise safety.
* Any medications, including St. John's wort, known to chronically alter drug absorption or elimination processes within 30 days prior to first dose administration.
* Subjects who smoke more than an average of 10 cigarettes per day.
* History of chronic alcohol or drug abuse within 12 months prior to screening.
* Subjects with ≥3 bowel movements per day.
* Any disorder which is not stable and could: Affect the safety of the subject throughout the trial; Influence the findings of the trial; Impede the subject's ability to complete the trial. Examples include but are not limited to cardiovascular, GI, hepatic, renal, neurological, musculoskeletal, infectious, endocrine, metabolic, haematological, immunological, and psychiatric disorders and major physical impairment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2019-01-22 (Actual); Primary Completion 2019-06-13 (Actual); Study Completion 2019-06-13 (Actual)

PRIMARY OUTCOMES:
Part 1. AUC0-∞ | Calculated using concentration data collected from predose to 48 hours postdose for each treatment period in Part 1
  AUC0-∞: Area under the plasma concentration-time curve from time 0 extrapolated to infinity
Part 1. Relative bioavailability (F-rel) | Calculated using concentration data collected from predose to 48 hours postdose for each treatment period in Part 1
  F-rel: AUC0 ∞ test formulations/AUC0-∞ reference formulation (derived from the statistical analysis of AUC0-∞)
Part 1. C-max | Calculated using concentration data collected from predose to 48 hours postdose for each treatment period in Part 1
  C-max: Maximum observed plasma concentration
Part 1. t-max | Calculated using concentration data collected from predose to 48 hours postdose for each treatment period in Part 1
  t-max: Time to reach maximum observed plasma concentration
Part 2. AUC0-∞ | Calculated using concentration data collected from predose to 72 hours postdose for each treatment period in Part 2
  AUC0-∞: Area under the plasma concentration-time curve from time 0 extrapolated to infinity
Part 2. Relative bioavailability (F-rel) | Calculated using concentration data collected from predose to 72 hours postdose for each treatment period in Part 2
  F-rel: AUC0 ∞ test formulations/AUC0-∞ reference formulation (derived from the statistical analysis of AUC0-∞)
Part 2. C-max | Calculated using concentration data collected from predose to 72 hours postdose for each treatment period in Part 2
  C-max: Maximum observed plasma concentration
Part 2. t-max | Calculated using concentration data collected from predose to 72 hours postdose for each treatment period in Part 2
  t-max: Time to reach maximum observed plasma concentration
Part 3. Number of GI-related AEs and number of subjects with GI-related AEs during the treatment period | From Day 1 (first dose) to Day 19 (end of treatment period) in Part 3
  AEs: adverse events; GI: gastrointestinal

SECONDARY OUTCOMES:
Part 1. Number of GI-related AEs and number of subjects with GI-related AEs during each combination of treatment and period. | 24 days (from first dose in first treatment period until end of last treatment period) in Part 1
  AEs: adverse events; GI: gastrointestinal
Part 1. Number of total AEs and number of subjects with AEs during each combination of treatment and period | 24 days (from first dose in first treatment period until end of last treatment period) in Part 1
  AEs: adverse events
Part 1. Number of subjects with systolic blood pressure in each of the following categories: 'normal', 'abnormal, not clinically significant', 'abnormal, clinically significant' | At screening and during each treatment period in Part 1: predose, 4 hours, 24 hours, and 48 hours postdose
  Normal: ≥90 and ≤140 mmHg. Clinical significance of abnormal values as judged by the investigator
Part 1. Number of subjects with diastolic blood pressure in each of the following categories: 'normal', 'abnormal, not clinically significant', 'abnormal, clinically significant' | At screening and during each treatment period in Part 1: predose, 4 hours, 24 hours, and 48 hours postdose
  Normal: ≥45 and ≤90 mmHg. Clinical significance of abnormal values as judged by the investigator
Part 1. Number of subjects with pulse rate in each of the following categories: 'normal', 'abnormal, not clinically significant', 'abnormal, clinically significant' | At screening and during each treatment period in Part 1: predose, 4 hours, 24 hours, and 48 hours postdose
  Normal: ≥40 and ≤100 beats/minute. Clinical significance of abnormal values as judged by the investigator
Part 1. Number of subjects with body temperature in each of the following categories: 'normal', 'abnormal, not clinically significant', 'abnormal, clinically significant' | At screening and during each treatment period in Part 1: predose, 4 hours, 24 hours, and 48 hours postdose
  Normal: ≥35 and ≤37.5°C. Clinical significance of abnormal values as judged by the investigator
Part 1. Number of subjects with PR interval in each of the following categories: 'normal', 'abnormal, not clinically significant', 'abnormal, clinically significant' | At screening, predose in Treatment period 1, and 48 hours postdose in Treatment period 3 in Part 1
  Normal: ≥120 and ≤220 msec. Clinical significance of abnormal values as judged by the investigator
Part 1. Number of subjects with QRS duration in each of the following categories: 'normal', 'abnormal, not clinically significant', 'abnormal, clinically significant' | At screening, predose in Treatment period 1, and 48 hours postdose in Treatment period 3 in Part 1
  Normal: ≤120 msec. Clinical significance of abnormal values as judged by the investigator
Part 1. Number of subjects with QTcF interval in each of the following categories: 'normal', 'abnormal, not clinically significant', 'abnormal, clinically significant' | At screening, predose in Treatment period 1, and 48 hours postdose in Treatment period 3 in Part 1
  QTcF: QT interval corrected for heart rate according to Fridericia's method. Normal: ≤450 msec for males and ≤470 msec for females. Clinical significance of abnormal values as judged by the investigator
Part 1. AUC0-t | Calculated using concentration data collected from predose to 48 hours postdose for each treatment period in Part 1
  AUC0-t: area under the plasma concentration time curve from time 0 to the time of last observed quantifiable concentration
Part 1. t1/2 | Calculated using concentration data collected from predose to 48 hours postdose for each treatment period in Part 1
  t1/2: apparent terminal half-life
Part 2. Number of GI-related AEs and number of subjects with GI-related AEs during each combination of treatment and period. | 28 days (from first dose in first treatment period until end of last treatment period) in Part 2
  AEs: adverse events; GI: gastrointestinal
Part 2. Number of total AEs and number of subjects with AEs during each combination of treatment and period | 28 days (from first dose in first treatment period until end of last treatment period) in Part 2
  AEs: adverse events
Part 2. Number of subjects with systolic blood pressure in each of the following categories: 'normal', 'abnormal, not clinically significant', 'abnormal, clinically significant' | At screening and during each treatment period in Part 2: predose, 4 hours, 24 hours, and 72 hours postdose
  Normal: ≥90 and ≤140 mmHg. Clinical significance of abnormal values as judged by the investigator
Part 2. Number of subjects with diastolic blood pressure in each of the following categories: 'normal', 'abnormal, not clinically significant', 'abnormal, clinically significant' | At screening and during each treatment period in Part 2: predose, 4 hours, 24 hours, and 72 hours postdose
  Normal: ≥45 and ≤90 mmHg. Clinical significance of abnormal values as judged by the investigator
Part 2. Number of subjects with pulse rate in each of the following categories: 'normal', 'abnormal, not clinically significant', 'abnormal, clinically significant' | At screening and during each treatment period in Part 2: predose, 4 hours, 24 hours, and 72 hours postdose
  Normal: ≥40 and ≤100 beats/minute. Clinical significance of abnormal values as judged by the investigator
Part 2. Number of subjects with body temperature in each of the following categories: 'normal', 'abnormal, not clinically significant', 'abnormal, clinically significant' | At screening and during each treatment period in Part 2: predose, 4 hours, 24 hours, and 72 hours postdose
  Normal: ≥35 and ≤37.5°C. Clinical significance of abnormal values as judged by the investigator
Part 2. Number of subjects with PR interval in each of the following categories: 'normal', 'abnormal, not clinically significant', 'abnormal, clinically significant' | At screening, predose in Treatment period 1, and 72 hours postdose in Treatment period 3 in Part 2
  Normal: ≥120 and ≤220 msec. Clinical significance of abnormal values as judged by the investigator
Part 2. Number of subjects with QRS duration in each of the following categories: 'normal', 'abnormal, not clinically significant', 'abnormal, clinically significant' | At screening, predose in Treatment period 1, and 72 hours postdose in Treatment period 3 in Part 2
  Normal: ≤120 msec. Clinical significance of abnormal values as judged by the investigator
Part 2. Number of subjects with QTcF interval in each of the following categories: 'normal', 'abnormal, not clinically significant', 'abnormal, clinically significant' | At screening, predose in Treatment period 1, and 72 hours postdose in Treatment period 3 in Part 2
  QTcF: QT interval corrected for heart rate according to Fridericia's method. Normal: ≤450 msec for males and ≤470 msec for females. Clinical significance of abnormal values as judged by the investigator
Part 2. AUC0-t | Calculated using concentration data collected from predose to 72 hours postdose for each treatment period in Part 2
  AUC0-t: area under the plasma concentration time curve from time 0 to the time of last observed quantifiable concentration
Part 2. t1/2 | Calculated using concentration data collected from predose to 72 hours postdose for each treatment period in Part 2
  t1/2: apparent terminal half-life
Part 3. AUC0-∞ | Calculated using concentration data collected from predose to 16 hours postdose on Day 17 in Part 3
  AUC0-∞: Area under the plasma concentration-time curve from time 0 extrapolated to infinity
Part 3. C-max | Calculated using concentration data collected from predose to 16 hours postdose on Day 17 in Part 3
  C-max: Maximum observed plasma concentration
Part 3. t-max | Calculated using concentration data collected from predose to 16 hours postdose on Day 17 in Part 3
  t-max: Time to reach maximum observed plasma concentration
Part 3. AUC0-t | Calculated using concentration data collected from predose to 16 hours postdose on Day 17 in Part 3
  AUC0-t: area under the plasma concentration time curve from time 0 to the time of last observed quantifiable concentration
Part 3. t1/2 | Calculated using concentration data collected from predose to 16 hours postdose on Day 17 in Part 3
  t1/2: apparent terminal half-life
Part 3. Number of total AEs and number of subjects with AEs during the treatment period | From Day 1 (first dose) to Day 19 (end of treatment period) in Part 3
  AEs: adverse events
Part 3. Number of subjects with systolic blood pressure in each of the following categories: 'normal', 'abnormal, not clinically significant', 'abnormal, clinically significant' | At screening and during the treatment period in Part 3: Days 1, 3, 5, 7, 9, and 11: predose and 4 hours postdose; Day 17: predose, 4 hours, and 12 hours postdose; Day 19 (=48 hours postdose)
  Normal: ≥90 and ≤140 mmHg. Clinical significance of abnormal values as judged by the investigator
Part 3. Number of subjects with diastolic blood pressure in each of the following categories: 'normal', 'abnormal, not clinically significant', 'abnormal, clinically significant' | At screening and during the treatment period in Part 3: Days 1, 3, 5, 7, 9, and 11: predose and 4 hours postdose; Day 17: predose, 4 hours, and 12 hours postdose; Day 19 (=48 hours postdose)
  Normal: ≥45 and ≤90 mmHg. Clinical significance of abnormal values as judged by the investigator
Part 3. Number of subjects with pulse rate in each of the following categories: 'normal', 'abnormal, not clinically significant', 'abnormal, clinically significant' | At screening and during the treatment period in Part 3: Days 1, 3, 5, 7, 9, and 11: predose and 4 hours postdose; Day 17: predose, 4 hours, and 12 hours postdose; Day 19 (=48 hours postdose)
  Normal: ≥40 and ≤100 beats/minute. Clinical significance of abnormal values as judged by the investigator
Part 3. Number of subjects with body temperature in each of the following categories: 'normal', 'abnormal, not clinically significant', 'abnormal, clinically significant' | At screening and during the treatment period in Part 3: Days 1, 3, 5, 7, 9, and 11: predose and 4 hours postdose; Day 17: predose, 4 hours, and 12 hours postdose; Day 19 (=48 hours postdose)
  Normal: ≥35 and ≤37.5°C. Clinical significance of abnormal values as judged by the investigator
Part 3. Number of subjects with PR interval in each of the following categories: 'normal', 'abnormal, not clinically significant', 'abnormal, clinically significant' | At screening and during the treatment period in Part 3: Day 1: predose and 4 hours postdose; Days 3, 5, 7, 9, 11, and 17: 4 hours postdose; Day 19 (=48 hours postdose)
  Normal: ≥120 and ≤220 msec. Clinical significance of abnormal values as judged by the investigator
Part 3. Number of subjects with QRS duration in each of the following categories: 'normal', 'abnormal, not clinically significant', 'abnormal, clinically significant' | At screening and during the treatment period in Part 3: Day 1: predose and 4 hours postdose; Days 3, 5, 7, 9, 11, and 17: 4 hours postdose; Day 19 (=48 hours postdose)
  Normal: ≤120 msec. Clinical significance of abnormal values as judged by the investigator
Part 3. Number of subjects with QTcF interval in each of the following categories: 'normal', 'abnormal, not clinically significant', 'abnormal, clinically significant' | At screening and during the treatment period in Part 3: Day 1: predose and 4 hours postdose; Days 3, 5, 7, 9, 11, and 17: 4 hours postdose; Day 19 (=48 hours postdose)
  QTcF: QT interval corrected for heart rate according to Fridericia's method. Normal: ≤450 msec for males and ≤470 msec for females. Clinical significance of abnormal values as judged by the investigator

CONTACTS AND LOCATIONS:
Overall Officials: Medical Expert, Study Director — LEO Pharma
Locations (1):
- LEO Pharma Investigational Site, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Data feasibility requests and research proposals are sent to disclosure@leo-pharma.com. If feasibility to share the data from a trial is granted, the ultimate decision is made by an external to the company board (Patient and Scientific Review Board). Data sharing is further subject to signed data sharing agreement. Data will be available in a closed environment for a specified period on time.
Supporting Information: Study Protocol, SAP, CSR
Access Criteria: External researchers with no commercial interest who provide scientifically sound research proposal
URL: http://www.leo-pharma.com/Home/Research-and-Development/Clinical-trial-disclosure/Access-to-patient-level-data.aspx